CLINICAL TRIAL: NCT03860467
Title: Epileptic Seizures in Intensive Care Units
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02361; me19Sutter
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Epileptic Seizure
Keywords: Status epilepticus; Electroencephalogram; Intensive Care Unit
MeSH Terms: conditions — Seizures; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of patient data — Patient data will be collected using the in-house digital patient record systems and the local digital electroencephalogram (EEG)-database

SUMMARY:
This retrospective observational cohort study is to assess and analyze clinical, electroencephalographic, laboratory, comorbidity, and treatment characteristics of Intensive care unit (ICU)-patients with epileptic seizures and to subsequently compare their characteristics with ICU-patients with status epilepticus (SE).

DETAILED DESCRIPTION:
The aim of this retrospective observational cohort study is to get further insight into adult patients with epileptic seizures in ICUs in an academic tertiary medical care center regarding frequency, clinical and electroencephalogram (EEG) characteristics, treatment, course and outcome. This data could help understanding the epidemiology (including risk factors, influence of EEG), and to guide management and improve outcomes of affected patients.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the ICU at the University Hospital Basel
* suffered from one or more epileptic seizures (detected clinically and/or by EEG) during their ICU-stay

Exclusion Criteria:

* patients with epileptic seizures transforming into Status epilepticus (SE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (i.e., ≥18 years of age) admitted to the ICUs at the University Hospital Basel that suffered from one or more epileptic seizures (detected clinically and/or by EEG) during their ICU-stay
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Frequency of epileptic seizures | between 01.01.2005 and 19.12.2018
  Frequency of all epileptic seizures in the ICU

SECONDARY OUTCOMES:
Number of epileptic seizures captured by EEG | between 01.01.2005 and 19.12.2018
  Number of epileptic seizures captured by EEG without overt clinical seizure presentation in the ICU
Number of epileptic seizures diagnosed on the basis of clinical symptoms alone | between 01.01.2005 and 19.12.2018
  Number of epileptic seizures diagnosed on the basis of clinical symptoms alone in the ICU
Length of epileptic seizure (time) | between 01.01.2005 and 19.12.2018
  Duration of epileptic seizure
Semiological feature of epileptic seizure (i.e. seizure types) | between 01.01.2005 and 19.12.2018
  Semiological feature of epileptic seizure (i.e. seizure types) emerging in ICU-patients

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, PD Dr. med, Principal Investigator — Clinic for Intensive Care Medicine, University Hospital Basel
Locations (1):
- Clinic for Intensive Care Medicine, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Wagner AS, Semmlack S, Frei A, Ruegg S, Marsch S, Sutter R. Seizures and risks for recurrence in critically ill patients: an observational cohort study. J Neurol. 2022 Aug;269(8):4185-4194. doi: 10.1007/s00415-022-11038-6. Epub 2022 Mar 2. PMID 35235003